CLINICAL TRIAL: NCT02999633
Title: Phase 2, Safety and Efficacy Study of Isatuximab, an Anti-CD38 Monoclonal Antibody, Administered by Intravenous (IV) Infusion in Patients With Relapsed or Refractory T-acute Lymphoblastic Leukemia (T-ALL) or T-lymphoblastic Lymphoma (T-LBL)
Brief Title: Safety and Efficacy of Isatuximab in Lymphoblastic Leukemia
Acronym: ISLAY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to an unsatisfactory benefit/risk ratio, as specified in & 14.8.1 of the protocol, Sanofi decided to stop enrollment and terminate ACT14596 prematurely
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT14596; 2016-002739-14 (EudraCT Number); U1111-1179-5294 (Other: UTN)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: T-cell Type Acute Leukemia-Precursor; T-lymphoblastic Lymphoma/Leukaemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — isatuximab; Dexamethasone; Acetaminophen; Ranitidine; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isatuximab (Experimental): Participants received intravenous administration of isatuximab at a dose of 20 milligrams/kilogram (mg/kg) at Day 1, 8, 15 and 22 of each Cycle (up to 2 treatment cycles, each cycle 28 days).
  Interventions: Drug: Isatuximab SAR650984; Drug: dexamethasone; Drug: acetaminophen; Drug: ranitidine; Drug: diphenhydramine

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form:solution Route of administration: intravenous
Drug: dexamethasone — Pharmaceutical form:pills Route of administration: oral
Drug: dexamethasone — Pharmaceutical form:solution Route of administration: intravenous
Drug: acetaminophen — Pharmaceutical form:pills Route of administration: oral
Drug: ranitidine — Pharmaceutical form:solution Route of administration: intravenous
Drug: diphenhydramine — Pharmaceutical form:solution Route of administration: intravenous

SUMMARY:
Primary Objective:

To evaluate the efficacy of isatuximab.

Secondary Objectives:

* To evaluate the safety profile of isatuximab.
* To evaluate the duration of response (DOR).
* To evaluate progression free survival (PFS) and overall survival (OS).
* To evaluate the pharmacokinetics (PK) of isatuximab in participants with T-ALL or T-LBL.
* To evaluate immunogenicity of isatuximab in participants with T-ALL or T-LBL.
* To assess minimal residual disease (MRD) and correlate it with clinical outcome.

DETAILED DESCRIPTION:
The study duration per participant included a 3-week screening period, an approximately 1 year of treatment period or until disease progression or discontinuation for any other reason, and a follow-up period of at least 30 days after the last investigational medicinal product administration.

ELIGIBILITY:
Inclusion criteria :

* Participants must had a known diagnosis of acute lymphoblastic leukemia (ALL) of T cell origin, including T-LBL and T-ALL with extramedullary involvement at relapse confirmed by biopsy.
* Participants must be previously treated for T-ALL or T-LBL and have relapsed or are refractory to most recent treatment. Participants in first relapse were be eligible regardless of the first remission duration.
* Participants must had been previously exposed to nelarabine in countries where this drug is available (unless due to a contraindication to its use or administrative issue).
* No more than 3 prior salvage therapies.

Exclusion criteria:

* Prior treatment with immunotherapy/investigational agents within 3 weeks, chemotherapy within 2 weeks of study treatment. Must have recovered from acute toxicity before first study treatment administration.
* Prior stem cell transplant within 4 months and/or evidence of active systemic Graft versus Host Disease and/or immunosuppressive therapy for Graft versus Host Disease within 1 week before the first study treatment administration.
* Clinical evidence of active central nervous system (CNS) leukemia.
* T-ALL with testicular involvement alone.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (17):
- United States (3):
  - Investigational Site Number 8400002, Atlanta, Georgia
  - Investigational Site Number 8400003, Hackensack, New Jersey
  - Investigational Site Number 8400001, Houston, Texas
- Investigational Site Number 2460001, Helsinki, Finland
- France (4):
  - Investigational Site Number 2500005, Nantes
  - Investigational Site Number 2500001, Paris
  - Investigational Site Number 2500004, Pessac
  - Investigational Site Number 2500002, Pierre-Bénite
- Hungary (3):
  - Investigational Site Number 3480001, Budapest
  - Investigational Site Number 3480003, Budapest
  - Investigational Site Number 3480002, Debrecen
- Italy (2):
  - Investigational Site Number 3800001, Bergamo
  - Investigational Site Number 3800004, Brescia
- Investigational Site Number 4400001, Vilnius, Lithuania
- Russia (3):
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430001, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Brillac C, Semiond D, Oprea C, Baruchel A, Zwaan CM, Nguyen L. Selection of isatuximab dosing regimen in pediatric patients with leukemia using population pharmacokinetics. Cancer Chemother Pharmacol. 2025 Dec 3;95(1):116. doi: 10.1007/s00280-025-04832-2. PMID 41331127
- [Derived] Wang A, Song Z, Zheng G, Nicolazzi C, Fromm JR, Shehu E, Srinivasan S, Chen X, Zhu C, Blondel MC, Adrian FJ. Evaluation of Preclinical Activity of Isatuximab in Patients with Acute Lymphoblastic Leukemia. Mol Cancer Ther. 2021 Oct;20(10):1916-1925. doi: 10.1158/1535-7163.MCT-21-0058. Epub 2021 Aug 10. PMID 34376579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 6 countries. A total of 16 participants were screened of those 2 participants failed screening: 1 participant for evidence of ongoing infection and 1 participant for not meeting the criterion for relapsed or refractory T-acute lymphoblastic leukemia (ALL)/T-lymphoblastic lymphoma (LBL).
Pre-assignment Details: The first participant was enrolled on 14 March 2017. A total of 14 participants were enrolled to receive isatuximab. The study was early terminated on 08 Nov 2017 due to an unsatisfactory benefit/risk ratio.
Period: Overall Study
Arm/Group | Isatuximab
Started | 14
Completed | 0
Not Completed | 14
Not completed — Adverse Event | 2
Not completed — Progressive disease | 12

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of isatuximab.
Groups:
- Isatuximab: Participants received intravenous administration of isatuximab at a dose of 20 mg/kg at Day 1, 8, 15 and 22 of each Cycle (up to 2 treatment cycles, each cycle 28 days).
Arm/Group | Isatuximab
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.36 (19.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response
Description: Objective response was defined as percentage of participants with complete response (CR) or with complete response with incomplete peripheral recovery (CRi) as per National Comprehensive Cancer Network (NCCN) guidelines. CR was defined as no circulating blasts or extramedullary disease, no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/central nervous system involvement, trilineage hematopoiesis and less than 5 percentage blasts, absolute neutrophil count (ANC) greater than 1000 per micro liter, platelets less than 100 000 per micro liter, no recurrence for 4 weeks. CRi meet all criteria for complete response except platelet count and/or ANC.
Time Frame: Baseline until disease progression or death (maximum duration: 12.1 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of isatuximab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Isatuximab
Number analyzed (Participants) | 14
percentage of participants | 0 [0 to 23.2]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as time (in days) from date of first response until date of first documented progressive disease (PD) or death (from any cause), whichever came first. Progressive disease as per NCCN guidelines was defined as increase of at least 25 percentage (%) in the absolute number of circulating or bone marrow blasts or development of extramedullary disease.
Time Frame: Baseline until disease progression or death (maximum duration: 12.1 weeks)
Population: The outcome measure was not analyzed due to lack of objective response. There was no specific additional data collected for the analysis of DOR as this outcome measure was to be derived using time point responses and death information that were collected and analyzed as part of primary and safety outcome measures, respectively.
Arm/Group | Isatuximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval (in days) from the date of first study drug administration to the date of first observation of PD or death due to any cause, whichever came first. PD as per NCCN guidelines was defined as increase of at least 25% in the absolute number of circulating or bone marrow blasts or development of extramedullary disease.
Time Frame: Baseline until disease progression or death (maximum duration: 12.1 weeks)
Population: This outcome measure was not analyzed because disease progression data were not collected.
Arm/Group | Isatuximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time interval from the date of first study drug administration to the date of death due to any cause.
Time Frame: Baseline until death (maximum duration: 12.1 weeks)
Population: This outcome measure was not analyzed because overall survival data were not collected.
Arm/Group | Isatuximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD)
Description: Presence of MRD was measured by sequencing and/or flow cytometry in participants achieving CR and CRi. CR was defined as no circulating blasts or extramedullary disease, no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/central nervous system involvement, trilineage hematopoiesis and less than 5 percentage blasts, ANC greater than 1000 per micro liter, platelets less than 100 000 per micro liter, no recurrence for 4 weeks. Complete response with incomplete blood count recovery meet all criteria for complete response except platelet count and/or ANC.
Time Frame: Baseline until death or study cut-off (maximum duration: 12.1 weeks)
Population: Data for this outcome measure was not collected and analyzed because no participant achieved CR or CRi.
Arm/Group | Isatuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug administration (up to maximum of 12.1 weeks)
Description: Reported Adverse events (AEs) are treatment emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from first study treatment administration until 30 days after the last administration of study treatment). Safety analysis set included all participants who received at least 1 dose of isatuximab.
Arm/Group | Isatuximab
All-Cause Mortality (participants affected / at risk) | 6/14
Serious Adverse Events (participants affected / at risk) | 10/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isatuximab (N=14)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Pericarditis Constrictive (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Disease Progression (General disorders) | 4 (4)
Device Related Infection (Infections and infestations) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1)
Periorbital Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pelvic Venous Thrombosis (Vascular disorders) | 1 (1)
Vein Collapse (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isatuximab (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (6)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1)
Pyelitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 8 (11)
Body Temperature Increased (Investigations) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle Oedema (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Facial Paralysis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02999633/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02999633/SAP_001.pdf